CLINICAL TRIAL: NCT01955005
Title: Pilot of My HealtheVet Training to Improve Co-Managed Care for Veterans
Brief Title: Use of the My HealtheVet for Health Information Sharing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 13-178
Record Dates: First submitted 2013-08-20; First posted 2013-10-07 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Illness
Keywords: Health Records, Personal; Delivery of healthcare; Consumer Participation; Internet
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- My HealtheVet Training (Experimental): Participants will be asked to watch an on-line training video, review written materials, and print a document containing health information from their My HealtheVet account.
  Interventions: Behavioral: My HealtheVet Training
- Internet Skills Training (Active Comparator): Participants will review written training materials to learn how to search the Internet for health information and how to decide which Internet sites have good quality information.
  Interventions: Other: Internet Skills Training

INTERVENTIONS:
Behavioral: My HealtheVet Training — Participants will be asked to watch an on-line training video, review written materials, and print a document containing health information from their My HealtheVet account.
  Arms: My HealtheVet Training
Other: Internet Skills Training — Participants will review written training materials to learn how to search the Internet for health information and how to decide which Internet sites have good quality information.
  Arms: Internet Skills Training

SUMMARY:
This study aims to conduct a pilot of an intervention to improve care coordination between VA and non-VA providers using the Department of Veteran's Affairs' (VA) personal health record, My HealtheVet (MHV). Participants will be randomized to receive either training on 1) how to use My HealtheVet to share VA health information or 2) training on how to how to search the Internet for health information and decide which Internet sites have good quality information. The investigators predict that Veterans who receive the My HealtheVet training will have fewer medication errors and duplication of services between the VA and outside providers.

DETAILED DESCRIPTION:
This study aims to conduct a pilot of an intervention to improve care coordination between VA and non-VA providers using the Department of Veteran's Affairs' (VA) personal health record, My HealtheVet (MHV). Background: The Blue Button feature of My HealtheVet allows Veterans to print out a comprehensive summary of their health that can be shared with non-VA providers. Dual use is common and has been associated with negative health outcomes including higher mortality. Preliminary data collected by the principal investigator in collaboration with the My HealtheVet Performance Evaluation workgroup shows that few Veterans enrolled in My HealtheVet use it to inform either VA or non-VA providers of their care. To remedy this, the principal investigator has developed an online video and companion paper-based training. This training will teach Veterans how to use the Blue Button feature and why it is important to share the print out with their non-VA provider. Methods: To participate, Veterans must have an upcoming non-VA provider appointment, be prescribed 5 or more medications, and be registered on My HealtheVet with a premium account. Participants will be randomized to receive either training on how to use the Blue Button or training on how to search for health information on the Internet and if that information is good quality. Veterans in both arms will receive training materials and phone support. After the non-VA provider visit, both the Veteran and the provider will be asked to indicate what occurred during the visit, including whether or not the Veteran gave the provider the Blue Button print out. Both Veterans and providers will also be asked to complete a 15-minute qualitative interview about their experience during the visit. Medical records of the non-VA provider visit will be obtained. Outcomes: The main outcome for the study is whether the patient provided the non-VA provider a copy of his or her health information printed from My HealtheVet. In addition, comparison between the VA and non-VA provider records will be conducted to test whether Veterans who completed the training had 1) better medication reconciliation between the VA and the non-VA provider and 2) fewer instances of therapeutic or laboratory duplication. The results of this pilot will be used to inform a larger randomized controlled trial of the training intervention.

ELIGIBILITY:
Inclusion Criteria:

* Upcoming Non-VA provider appointment
* Take 5 or more prescribed medications
* Have or obtain a My HealtheVet premium account
* Access to computer, printer, & Internet to complete study protocol

Exclusion Criteria:

* No non-VA provider or upcoming appointment
* Less than 5 medications
* No premium MHV account

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Turvey, PhD MS, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | My HealtheVet Training | Internet Skills Training
Started | 30 | 30
Completed | 27 | 25
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Population: Veterans with a diagnosis of at least one chronic health condition taking 5 or more medications who have both a VA and a non-VA provider.
Groups:
- Total: Total of all reporting groups
Arm/Group | My HealtheVet Training | Internet Skills Training | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (6.0) | 68.5 (6.4) | 68.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 25 | 21 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 26 | 22 | 48
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Brought Their VA Information From My HealtheVet to Their Visit With Their Non-VA Provider
Description: The primary outcome is whether or not the veteran brings their VA information from My HealtheVet to their visit with their non-VA provider. Providers will be asked to complete a form during the appointment where assessment of sharing this information is embedded in a checklist of possible visit activities. Participants will also if they provided this information to the provider in the event the provider opts to not return the form.
Time Frame: Within 1-2 week of non-VA provider visit
Population: This outcome was collected from the provider completed questionnaire. The reduced sample size is due to the response rate for the My Healthe Vet training group providers (74%) and the Internet Skills Training group (52%).
Measure: Number; unit: Percentage of Participants
Arm/Group | My HealtheVet Training | Internet Skills Training
Number analyzed (Participants) | 21 | 12
Percentage of Participants | 90 | 6
Statistical Analysis 1: Comparison: My HealtheVet Training vs Internet Skills Training; This was a 2x2 comparison using Fisher's exact due to low expected cell count. Fisher's exact p<0.001; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Proportion of Total Number of Unique Medications Discrepant Between VA and Non-VA Medication Lists
Description: A medication discrepancy metric was be calculated by comparing the current VA medication list with the non-VA provider medication list to determine the total number of distinct medications. The number of discrepant medications between these lists is the numerator and is divided by the total number of distinct medications on both lists combined. This will yield a range of scores between score between 0 and 1, with 1 indicating perfect agreement between the two lists.
Time Frame: Typically within 1 month of non-VA provider visit
Population: Medication reconciliation was based on Medical Record Review, therefore there was better representation of the entire sample. 2 Veterans were not included in the Internet Skills Training group because the medical records sent from the Non-VA provider were not adequate to determine an accurate medication list.
Measure: Mean (Standard Deviation); unit: proportion of medications discrepant
Arm/Group | My HealtheVet Training | Internet Skills Training
Number analyzed (Participants) | 27 | 23
proportion of medications discrepant | 0.49 (0.25) | 0.44 (0.23)
Statistical Analysis 1: Comparison: My HealtheVet Training vs Internet Skills Training; Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney); Z score = 568.5

3. Secondary Outcome: Proportion of Participants Who Received One or More Duplicate Laboratory Tests in the Non-VA Provider Visit.
Description: Therapeutic duplication will be defined as concurrent use of more than one medication from the same therapeutic class. For laboratory duplication, we will review non-VA and VA medical records 6 months prior to the non-VA provider visit. Each patient will be assigned a dichotomous indicator for whether they received therapeutic duplication and/or laboratory duplication during their non-VA provider visit
Time Frame: Typically within 1 month of non-VA provider visit
Population: Some veterans had their laboratories drawn prior to the medical visit and were therefore excluded from this analysis.
Measure: Number; unit: proportion of participants
Arm/Group | My HealtheVet Training | Internet Skills Training
Number analyzed (Participants) | 20 | 22
proportion of participants | 0 | 27
Statistical Analysis 1: Comparison: My HealtheVet Training vs Internet Skills Training; Test type: Superiority or Other; p = 0.02, Fisher's Exact; Table Probability = 0.0142

ADVERSE EVENTS:
Time Frame: One Year
Description: This is a low risk study. The only potential adverse event was inadvertent confidentiality breech.
Arm/Group | My HealtheVet Training | Internet Skills Training
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes